CLINICAL TRIAL: NCT05324605
Title: Personalized 3D Virtual and Printed Model Versus Conventional Images for the Education of the Treatment Planning in Intracranial Aneurysm Surgeries.
Brief Title: Personalized Treatment Planning in Intracranial Aneurysm Surgeries.
Acronym: 3 D
Status: Completed | Type: Observational
Sponsor: Prof. Dr. med. Serge Marbacher (Other)
Collaborators: Kantonsspital Aarau (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Serge Marbacher, Prof. Dr. med., Kantonsspital Aarau
Organization: Kantonsspital Aarau (Other)
Other Study IDs: 3 D
Record Dates: First submitted 2022-04-06; First posted 2022-04-12 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Aneurysm Cerebral
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Questionnaire and use of 3 D tools — Resulting computer tomography(CT) results are transferred to a 3 D projection. Patients will be asked to wear 3 D glasses to be able visualizing the diagnosed vascular pathology. The physician will explain the disaese and treatment. The patient is ask to fill out a questionnaire post 3D consulting

SUMMARY:
Patients who will undergo a intracranial aneurysm (IA) surgery are educated concerning their disease and the surgical procedure.The objective of this study is to explore the advantages of conventional, virtual reality and 3D stereolithographic models for patient and resident education in the treatment of lAs.

DETAILED DESCRIPTION:
Patient understanding of their medical condition and treatment satisfaction has gained increasing attention in medicine. As for neurosurgical conditions however, the treatment plan is often difficult for patients to comprehend, with many of them having an inaccurate understanding of the involved anatomy.

Novel technologies therefore may play a role in facilitating patient education. In particular, conventional 2D images makes it sometimes difficult for surgeons to inform their patients about the planned intervention and potential complications. This is why new modalities have been developed for patient information and may have further an impact on resident education to better estimate the treatment plan and potential complication. For the latter, given that intracranial aneurysms (lAs) are increasingly treated via endovascular methods, training opportunities are reduced and understanding of the vascular anatomy can become difficult.

The objective of this study is to explore the advantages of conventional, virtual reality and 3D stereolithographic models for patient and resident education in the treatment of lAs.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective surgery for non-ruptured IA during the study period will be considered for inclusion. Patients are included if they are at least 18 years old and are able to give informed consent and signed the informed consent form.

Exclusion Criteria:

* Patients with ruptured or mycotic IA are not considered. Furthermore, patients elected for IA surgery that are younger than 18 years old, as well as patients who are unable to give informed consent (e.g. neurological impairments) will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are patient with a age >18 years, diagnosed with a intracranial aneurysma , requiring surgery. The eligibility is evaluated and prior surgery, preoperative assessment by CTA and 3D-DSA have been performed. After screening a non routine consultation with the 3 D method visualization is scheduled. Finally, patients will be scheduled for surgery according to our standard procedure.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
accuracy of the planned intervention and clip placement. | 6 months post interventional
  Assessment of the 3D models regarding the accuracy of the planned intervention. In specific the following surgical steps are evaluated and assessed during aneurysm clipping and compared to the ideal preoperative forecast based on the 3D model (GRF_clip anticipation): Temporary clips: (1) number of temporary clips; (2) left- or right-handed application; (3) position on parent artery; (4) length of the clip; (5) shape of the clip. Permanent clips: (6) number of permanent clips; (7) left- or right-handed application; (8) length of the clip; (9) shape of the clip.

SECONDARY OUTCOMES:
patient education | 6 months post interventional
  Assessment of ischemia (large and perforating artery compromise), time of temporary clip occlusion, morbidity, clinical outcome., To investigate the impact of personalized 3D printed model on patient information before surgery, study participants will be presented with their individual 3D printed model and a questionaire to analze an improvement in their understanding of basic anatomy, the planned surgical procedure, and understanding the complications related to the surgery will be assessed (GRF_patient satisfaction).
  To further determine if 3D printed models can be used to improve intraoperative pattern recognition and be a valuable adjunct in neurosurgical resident education, a comparison of conventional imaging with CT-scan, 3D-RA, 3D model will be assessed (GRF_resident education).

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Aarau AG, Aarau, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vlak MH, Algra A, Brandenburg R, Rinkel GJ. Prevalence of unruptured intracranial aneurysms, with emphasis on sex, age, comorbidity, country, and time period: a systematic review and meta-analysis. Lancet Neurol. 2011 Jul;10(7):626-36. doi: 10.1016/S1474-4422(11)70109-0. PMID 21641282
- [Background] Andereggen L, Gralla J, Andres RH, Weber S, Schroth G, Beck J, Widmer HR, Reinert M, Raabe A, Peterhans M. Stereolithographic models in the interdisciplinary planning of treatment for complex intracranial aneurysms. Acta Neurochir (Wien). 2016 Sep;158(9):1711-20. doi: 10.1007/s00701-016-2892-3. Epub 2016 Jul 14. PMID 27416860
- [Background] Kimura T, Morita A, Nishimura K, Aiyama H, Itoh H, Fukaya S, Sora S, Ochiai C. Simulation of and training for cerebral aneurysm clipping with 3-dimensional models. Neurosurgery. 2009 Oct;65(4):719-25; discussion 725-6. doi: 10.1227/01.NEU.0000354350.88899.07. PMID 19834377
- [Background] Russin J, Babiker H, Ryan J, Rangel-Castilla L, Frakes D, Nakaji P. Computational Fluid Dynamics to Evaluate the Management of a Giant Internal Carotid Artery Aneurysm. World Neurosurg. 2015 Jun;83(6):1057-65. doi: 10.1016/j.wneu.2014.12.038. Epub 2014 Dec 22. PMID 25541083
- [Background] Slichter SJ. Platelet transfusion therapy. Hematol Oncol Clin North Am. 1990 Feb;4(1):291-311. PMID 2179213
- [Background] Tanabe J, Ishikawa T, Moroi J, Sakata Y, Hadeishi H. Impact of Right-Sided Aneurysm, Rupture Status, and Size of Aneurysm on Perforator Infarction Following Microsurgical Clipping of Posterior Communicating Artery Aneurysms with a Distal Transsylvian Approach. World Neurosurg. 2018 Mar;111:e905-e911. doi: 10.1016/j.wneu.2018.01.002. Epub 2018 Jan 8. PMID 29325945
- [Background] Roszelle BN, Babiker MH, Hafner W, Gonzalez LF, Albuquerque FC, Frakes DH. In vitro and in silico study of intracranial stent treatments for cerebral aneurysms: effects on perforating vessel flows. J Neurointerv Surg. 2013 Jul;5(4):354-60. doi: 10.1136/neurintsurg-2012-010322. Epub 2012 Jun 26. PMID 22735859